CLINICAL TRIAL: NCT03645785
Title: Variation in Urine Electrolytes, pH and Specific Gravity Throughout the Day and the Effect of Increased Fluid Intake on Intra-Day Urine Composition
Brief Title: Variation in Urine Electrolytes, pH and Specific Gravity Throughout the Day
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adam Howe, MD (Other)
Collaborators: Labcorp Corporation of America Holdings, Inc (Industry)
Responsible Party: Sponsor-Investigator, Adam Howe, MD, Assistant Professor of Surgery, Albany Medical College
Organization: Albany Medical College (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: AMC5086
Record Dates: First submitted 2018-05-30; First posted 2018-08-24 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: All subjects will collect 4 urine samples on Day1 and Day 4. On day 2, 3 and 4 all subjects will drink a bottle of water with True Lemon and collect another 4 urine samples on day 4
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Diet/Drinking (Active Comparator): Baseline diet and drinking patterns for patients. This is the pre-intervention baseline for cross-over analysis
  Interventions: Dietary Supplement: Normal fluid intake without true lemon
- Increased fluid Intake and Citrate Supplementation (Experimental): Patients will increase fluid (with goal to double their baseline) and further take a citrate supplement in the form of True Lemon (citric acid).
  Interventions: Dietary Supplement: Double fluid intake plus 3 bottles of water with True Lemon

INTERVENTIONS:
Dietary Supplement: Normal fluid intake without true lemon — 16.9oz water with True Lemon
  Arms: Normal Diet/Drinking
Dietary Supplement: Double fluid intake plus 3 bottles of water with True Lemon — No intervention
  Arms: Increased fluid Intake and Citrate Supplementation

SUMMARY:
This study is a prospective study looking at healthy adults who will have urine collected at 4 set times throughout the course of the day. On Day 2, 3, and 4 subjects will drink a bottle of water containing True lemon and on days 2 and 3 double the amount of fluid intake from Day 1. On day 4 the subject will collect urine samples at 4 set times throughout the day. The pH of all of the urine samples will be checked with a urine dipstick and the samples will be sent to Litholink Lab for electrolyte composition analysis.

DETAILED DESCRIPTION:
20 subjects will be recruited and consented in the Urology Clinic office. Subjects will complete a questionnaire asking about weight, height, history of kidney stones, whether they are on any diuretics, medications that alter urine chemistries, or special diets. BMI will be calculated. Day 1 will begin at 5p.m. on the day before first morning void is collected. The subjects will collect a spot urine sample on the first void at home, then at 9-10AM, 1-2 PM and 4-5PM. They will be provided 4 sterile urine cups labeled for the different timed collection marked at the 20-30 ml line to indicate how much urine should be collected. Subjects will be instructed to refrigerate their first voids.The 2nd, 3rd and 4th void samples will be collected in the office during the designated times, and given to study personnel. The subjects will record the time of each void, the time given to the study representative, the times they eat, and their approximate fluid intake on the provided diaries. Subjects will be asked not to void outside of the timed collections. If they do void outside of these times, they will be asked to record the extra times that they void.

On Day 2, 3, and 4 the subject will drink a bottle of water with True Lemon after 5pm. On days 3 and 4 the subjects will double their fluid intake using Day 1 as a guide. On Day 4 the subjects will collect 4 urine samples as previously described for Day1. They will be instructed to mix 1 packet of True lemon in one 16.9oz (500 mL) bottle of Poland Spring. All True Lemon packets (True Citrus, 11501 Pocomoke Court Suite D, Baltimore, MD 21220). and Poland Spring (Nestle Waters North America) bottles will be provided to subjects by the research study team.

UA dipsticks will be used in office to evaluate for pH and specific gravity. Samples will also be sent to lab for evaluation of chemical composition of creatinine, citrate, and calcium. Electrolytes will be indexed against creatinine to evaluate their concentrations without having a 24-hour void volume amount A sample of citrate-Poland Spring will be sent to Litholink for analysis of Calcium and Citrate for reference.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects

Exclusion Criteria:

* Subjects taking diuretics
* Subjects who have known kidney disease
* Subjects with history of known nephrolithiasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Howe, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical College, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheungpasitporn W, Rossetti S, Friend K, Erickson SB, Lieske JC. Treatment effect, adherence, and safety of high fluid intake for the prevention of incident and recurrent kidney stones: a systematic review and meta-analysis. J Nephrol. 2016 Apr;29(2):211-219. doi: 10.1007/s40620-015-0210-4. Epub 2015 May 29. PMID 26022722
- [Background] Lotan Y, Antonelli J, Jimenez IB, Gharbi H, Herring R, Beaver A, Dennis A, Von Merveldt D, Carter S, Cohen A, Poindexter J, Moe OW, Pearle MS. The kidney stone and increased water intake trial in steel workers: results from a pilot study. Urolithiasis. 2017 Apr;45(2):177-183. doi: 10.1007/s00240-016-0892-7. Epub 2016 May 26. PMID 27228999
- [Background] Scales CD Jr, Smith AC, Hanley JM, Saigal CS; Urologic Diseases in America Project. Prevalence of kidney stones in the United States. Eur Urol. 2012 Jul;62(1):160-5. doi: 10.1016/j.eururo.2012.03.052. Epub 2012 Mar 31. PMID 22498635
- [Background] Pearle MS, Goldfarb DS, Assimos DG, Curhan G, Denu-Ciocca CJ, Matlaga BR, Monga M, Penniston KL, Preminger GM, Turk TM, White JR; American Urological Assocation. Medical management of kidney stones: AUA guideline. J Urol. 2014 Aug;192(2):316-24. doi: 10.1016/j.juro.2014.05.006. Epub 2014 May 20. PMID 24857648
- [Background] Hong YH, Dublin N, Razack AH, Mohd MA, Husain R. Twenty-four hour and spot urine metabolic evaluations: correlations versus agreements. Urology. 2010 Jun;75(6):1294-8. doi: 10.1016/j.urology.2009.08.061. Epub 2009 Nov 14. PMID 19914693
- [Background] Omar M, Sarkissian C, Jianbo L, Calle J, Monga M. Dipstick Spot urine pH does not accurately represent 24 hour urine PH measured by an electrode. Int Braz J Urol. 2016 May-Jun;42(3):546-9. doi: 10.1590/S1677-5538.IBJU.2015.0071. PMID 27286119
- [Background] Strohmaier WL, Hoelz KJ, Bichler KH. Spot urine samples for the metabolic evaluation of urolithiasis patients. Eur Urol. 1997;32(3):294-300. PMID 9358216
- [Background] Fenton TR, Eliasziw M, Lyon AW, Tough SC, Brown JP, Hanley DA. Low 5-year stability of within-patient ion excretion and urine pH in fasting-morning-urine specimens. Nutr Res. 2009 May;29(5):320-6. doi: 10.1016/j.nutres.2009.04.005. PMID 19555813
- [Background] Matsushita K, Tanikawa K. Significance of the calcium to creatinine concentration ratio of a single-voided urine specimen in patients with hypercalciuric urolithiasis. Tokai J Exp Clin Med. 1987 Sep;12(3):167-71. PMID 3454077
- [Background] Utsch B, Klaus G. Urinalysis in children and adolescents. Dtsch Arztebl Int. 2014 Sep 12;111(37):617-25; quiz 626. doi: 10.3238/arztebl.2014.0617. PMID 25283761
- [Background] Simerville JA, Maxted WC, Pahira JJ. Urinalysis: a comprehensive review. Am Fam Physician. 2005 Mar 15;71(6):1153-62. PMID 15791892
- [Background] Hardy PE. Urinalysis interpretation. Neonatal Netw. 2010 Jan-Feb;29(1):45-9. doi: 10.1891/0730-0832.29.1.45. No abstract available. PMID 20085877
- [Background] Yi JH, Shin HJ, Kim SM, Han SW, Kim HJ, Oh MS. Does the exposure of urine samples to air affect diagnostic tests for urine acidification? Clin J Am Soc Nephrol. 2012 Aug;7(8):1211-6. doi: 10.2215/CJN.03230312. Epub 2012 Jun 14. PMID 22700881
- [Background] Taylor EN, Curhan GC. Body size and 24-hour urine composition. Am J Kidney Dis. 2006 Dec;48(6):905-15. doi: 10.1053/j.ajkd.2006.09.004. PMID 17162145
- [Background] Curhan GC, Willett WC, Speizer FE, Stampfer MJ. Twenty-four-hour urine chemistries and the risk of kidney stones among women and men. Kidney Int. 2001 Jun;59(6):2290-8. doi: 10.1046/j.1523-1755.2001.00746.x. PMID 11380833
- [Background] Ahmed AI, Baz H, Lotfy S. Urinalysis: The Automated Versus Manual Techniques; Is It Time To Change? Clin Lab. 2016;62(1-2):49-56. doi: 10.7754/clin.lab.2015.150520. PMID 27012033
- [Background] LaRocco MT, Franek J, Leibach EK, Weissfeld AS, Kraft CS, Sautter RL, Baselski V, Rodahl D, Peterson EJ, Cornish NE. Effectiveness of Preanalytic Practices on Contamination and Diagnostic Accuracy of Urine Cultures: a Laboratory Medicine Best Practices Systematic Review and Meta-analysis. Clin Microbiol Rev. 2016 Jan;29(1):105-47. doi: 10.1128/CMR.00030-15. PMID 26598386
- [Background] Lifshitz E, Kramer L. Outpatient urine culture: does collection technique matter? Arch Intern Med. 2000 Sep 11;160(16):2537-40. doi: 10.1001/archinte.160.16.2537. PMID 10979067
- [Background] Morimoto M, Yanai H, Shukuya K, Chiba H, Kobayashi K, Matsuno K. Effects of midstream collection and the menstrual cycle on urine particles and dipstick urinalysis among healthy females. Clin Chem. 2003 Jan;49(1):188-90. doi: 10.1373/49.1.188. No abstract available. PMID 12507982
- [Background] Worcester EM, Coe FL, Evan AP, Bergsland KJ, Parks JH, Willis LR, Clark DL, Gillen DL. Evidence for increased postprandial distal nephron calcium delivery in hypercalciuric stone-forming patients. Am J Physiol Renal Physiol. 2008 Nov;295(5):F1286-94. doi: 10.1152/ajprenal.90404.2008. Epub 2008 Aug 20. PMID 18715937
- [Background] Desai RA, Assimos DG. Accuracy of urinary dipstick testing for pH manipulation therapy. J Endourol. 2008 Jun;22(6):1367-70. doi: 10.1089/end.2008.0053. PMID 18578664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from Albany Medical Center Urology clinic. A total of 23 participants were recruited
Pre-assignment Details: 23 patients were enrolled, but 3 had to be excluded based on study exclusion criteria.
  3 patients had a history of nephrolithiasis.
Groups:
- Non-Stone Forming: All 23 patients completed both interventions, and were used as their own control for baseline vs increased fluid/citrate intake comparisons in this cross over study.
  The same cohort underwent the following 2 periods, and all participants competed both
  Period 1: Normal drinking habits and diet. This was for a total of 24 hours (i.e. Day 1). Urine was collected throughout day 1
  Period 2: Increased fluid intake and citrate supplement (I.e. day 2-4). Participants all were encouraged to double their baseline fluid intake compared to day 1, and drink 1 bottle of Poland Spring 16.9oz with 1 packet of True lemon per day. Urine was collected throughout day 4.
Period: Day 1 (Normal Fluid Intake and Diet)
Arm/Group | Non-Stone Forming
Started | 23
Completed | 23
Not Completed | 0
Period: Day 2-4 (Double Fluid and Add Citrate)
Arm/Group | Non-Stone Forming
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 3 patients were excluded due to history of stones in the analysis
Groups:
- Non-Stone Forming Cohort: All 23 patients completed both interventions, and were used as their own control for baseline vs increased fluid/citrate intake comparisons in this cross over study.
  The same cohort underwent the following 2 periods, and all participants competed both
  Period 1: Normal drinking habits and diet. This was for a total of 24 hours (i.e. Day 1). Urine was collected throughout day 1
  Period 2: Increased fluid intake and citrate supplement (I.e. day 2-4). Participants all were encouraged to double their baseline fluid intake compared to day 1, and drink 1 bottle of Poland Spring 16.9oz with 1 packet of True lemon per day. Urine was collected throughout day 4.
Arm/Group | Non-Stone Forming Cohort
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants] — We did not measure age in this study. Only patients above the age of 18 were included, but this was screened for prior to recruitment.
  Participants
    Age >/= 18 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Full Range); unit: kg/m^2] | 25.9 [19.4 to 44.9]
Use of Vitamins [Count of Participants; unit: Participants] | 8
Diet [Count of Participants; unit: Participants]
  Vegetarians | 2
  Clean | 1
  Gluten Free | 1

OUTCOME MEASURES:

1. Primary Outcome: Citrate/Creatinine Ratio
Description: Citrate/Cr at 4 voids throughout the day. Pre = baseline fluid intake; Post = increased fluid and citrate supplementation
Time Frame: Day 1 (first void, 9-10 am, 1-2 pm and 5 pm) and Day 4 (first void, 9-10 am, 1-2 pm and 5 pm)
Population: Each participant had urine collected at each time listed: Day 1 (first void, 9-10 am, 1-2 pm and 5 pm) and Day 4 (first void, 9-10 am, 1-2 pm and 5 pm). Data was collected on the Citrate/Creatinine Ratio at each time period void. Thus, at each time of day, there was an N equivalent to the number of voids across all entire 20 participant cohort. Since it was the same participant providing the void at the different times, the sum of participants does not add to the n in the study population (20).
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- 5pm Void Post: increased fluid intake cohort 5p.m void
- 5p.m. Pre: normal fluid intake 5 p.m void
- 1-2 pm Post; 9-10AM Post: void time post intervention
- 1-2pm Void Pre; 9-10AM Pre: void time pre intervention
- First Void Pre: pre intervention, first void
- First Void Post: post intervention post void
Arm/Group | 5pm Void Post | 5p.m. Pre | 1-2 pm Post | 1-2pm Void Pre | 9-10AM Post | 9-10AM Pre | First Void Pre | First Void Post
Number analyzed (Participants) | 19 | 20 | 19 | 20 | 20 | 20 | 20 | 20
ratio | 0.658644 (0.429258801) | 0.584115 (0.393029128) | 0.562886 (0.309518524) | 0.540394 (0.332082046) | 0.490685 (0.246362039) | 0.441938 (0.209042617) | 0.423415 (0.22046721) | 0.404892 (0.248163828)

2. Primary Outcome: Calcium / Creatinine
Description: Ca/Cr at 4 voids throughout the day. Pre = baseline fluid intake; Post = increased fluid and citrate supplementation
Time Frame: Day 1 (first void, 9-10 am, 1-2 pm and 5 pm) and Day 4 (first void, 9-10 am, 1-2 pm and 5 pm)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 5pm Void Post | 5p.m. Pre | 1-2 pm Post | 1-2pm Void Pre | 9-10AM Post | 9-10AM Pre | First Void Pre | First Void Post
Number analyzed (Participants) | 19 | 20 | 19 | 20 | 20 | 20 | 20 | 20
Ratio | 0.162234 (0.114914139) | 0.161287 (0.166305391) | 0.137398 (0.1035436) | 0.140431 (0.153463692) | 0.126269 (0.097422413) | 0.111446 (0.072068182) | 0.160932 (0.111594912) | 0.142987 (0.108493894)

3. Primary Outcome: pH
Description: pH at 4 voids throughout the day. Pre = baseline fluid intake; Post
Time Frame: Day 1 (first void, 9-10 am, 1-2 pm and 5 pm) and Day 4 (first void, 9-10 am, 1-2 pm and 5 pm)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | 5pm Void Post | 5p.m. Pre | 1-2 pm Post | 1-2pm Void Pre | 9-10AM Post | 9-10AM Pre | First Void Pre | First Void Post
Number analyzed (Participants) | 19 | 20 | 19 | 20 | 20 | 20 | 20 | 20
pH | 6.52770 (0.479508661) | 6.32645 (0.666506167) | 6.34060 (0.621006253) | 6.37845 (0.616991723) | 6.43430 (0.729245327) | 6.24125 (0.70866872) | 6.08345 (0.47842631) | 6.01865 (0.477511011)

4. Primary Outcome: Specific Gravity (SG)
Description: SG at 4 voids throughout the day. Pre = baseline fluid intake; Post
Time Frame: Day 1 (first void, 9-10 am, 1-2 pm and 5 pm) and Day 4 (first void, 9-10 am, 1-2 pm and 5 pm)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/mL
Arm/Group | 5pm Void Post | 5p.m. Pre | 1-2 pm Post | 1-2pm Void Pre | 9-10AM Post | 9-10AM Pre | First Void Pre | First Void Post
Number analyzed (Participants) | 19 | 20 | 20 | 20 | 20 | 20 | 20 | 20
g/mL | 1.01725 (0.003851644) | 1.01525 (0.005773503) | 1.01725 (0.005799975) | 1.01850 (0.005745131) | 1.01950 (0.003906066) | 1.02051 (0.005058298) | 1.02000 (0.004552929) | 1.01825 (0.004537426)

5. Primary Outcome: Total Fluid Intake
Time Frame: Over 4 day study period
Population: Each participant completed the study, having their total fluid intake measured on each day. Thus, the overall number of participants does not add to the study total (n=20) as each participant
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Day 1: (Baseline)
- Day 2; Day 3; Day 4: (Increased Fluid + Citrate)
Arm/Group | Day 1 | Day 2 | Day 3 | Day 4
Number analyzed (Participants) | 20 | 20 | 20 | 20
mL | 2416.854 (1033) | 2625.093 (663.8) | 3116.562 (1308) | 3396.781 (1312)

ADVERSE EVENTS:
Time Frame: 4 days.
Groups:
- Normal Drinking Habits; Increased Fluid Intake and Citrate Supplementation: There were no adverse effects noted. Data was collected for the 4 day study period.
Arm/Group | Normal Drinking Habits | Increased Fluid Intake and Citrate Supplementation
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
Small number of study participants. Perhaps because we required participants to submit four fresh urine samples promptly throughout two separate days, 3 days apart, recruitment for the study was difficult. No nighttime urine collections. Further, we did not collect 24 hour urine samples simultaneously with the spot urines. One further limitation is that this looked at normal control patients only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT03645785/Prot_SAP_000.pdf